CLINICAL TRIAL: NCT02015312
Title: A Randomised Trial for the Treatment of Cardiac AMyloid Light-chain Amyloidosis With the Green Tea Compound Epigallocatechin-3-gallate (TAME-AL)
Brief Title: A Trial for the Treatment of Cardiac AL-Amyloidosis With the Green Tea Compound Epigallocatechin-3-gallate (TAME-AL)
Acronym: TAME-AL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florian Michel (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Florian Michel, Study Coordinator, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAME-AL; 2012-004520-38 (EudraCT Number)
Record Dates: First submitted 2013-11-18; First posted 2013-12-19 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Light Chain (AL) Amyloidosis; Cardiac Involvement
Keywords: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — epigallocatechin gallate; epigallocatechin-3-(3''-O-methyl)gallate; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epigallocatechin-3-gallate (EGCG) (Experimental): EGCG 400 mg/d p.o. for 3 months; 800 mg/d p.o. for 3 months, 1200 mg/d p.o. for 6 months
  Interventions: Drug: Epigallocatechin-3-gallate (EGCG)
- Placebo (Placebo Comparator): capsules
  Dose:
  400 mg/d for 3 months; 800 mg/d for 3 months, 1200 mg/d for 6 months Route of administration: p.o. Treatment duration: 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epigallocatechin-3-gallate (EGCG) — Pharmaceutical formulation: capsules
  Dose:
  400 mg/d for 3 months; 800 mg/d for 3 months, 1200 mg/d for 6 months Route of administration: p.o. Treatment duration: 12 months
  Other Names: Epigallocatechin gallate; EGCG; Epigallocatechin 3-gallate; Tea catechin; Epigallocatechin-3-gallate
  Arms: Epigallocatechin-3-gallate (EGCG)
Drug: Placebo — Pharmaceutical formulation: capsules
  Dose:
  400 mg/d for 3 months; 800 mg/d for 3 months, 1200 mg/d for 6 months Route of administration: p.o. Treatment duration: 12 months
  Other Names: Mannitol 99.5% + highly dispersed silicon dioxide 0.5%
  Arms: Placebo

SUMMARY:
Efficacy and safety of epigallocatechin-3-gallate (EGCG) in patients with cardiac amyloid light-chain (AL) amyloidosis. Evaluation of clinical efficacy of EGCG intake using a pretest posttest comparison of left ventricular amyloid mass (g/m2) measured by cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven systemic AL amyloidosis.
* Cardiac involvement with septum thickness more than 12 mm (without other causes as published by Gertz et al., hypertension or other potential causes of left ventricular hypertrophy)
* Previously treated with chemotherapy, induced at least a very good partial remission of the underlying monoclonal plasma cell or B cell disorder.
* GPT and GOT less than 3-times ULN.
* Life expectancy more than 12 month.
* Ability of subject to understand character and individual consequences of the clinical trail.
* Written informed consent.
* For women with childbearing potential and men, adequate contraception.

Exclusion Criteria:

* Age less than 18 years.
* Concomitant multiple myeloma stage 2 and 3 (Salmon and Durie)
* Concurrent chemotherapy necessary
* Time to last chemotherapy more than 6 months.
* Chronic liver disease, Bilirubin over 1,5 mg/dl
* Not able to visit Amyloidosis Clinic in Heidelberg every 3 months.
* History of hypersensitivity to the investigational product or to any substance with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other clinical trials or observation period of competing trials, respectively.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-04; Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
compare the 12 month change in left ventricular mass | 12 month
  The primary analysis to compare the 12 month change in left ventricular mass between the two treatment arms will be performed by a one-sided two-sample t test at a significance level of 0.025.

SECONDARY OUTCOMES:
Change in Quality of Life | baseline, 12 month
  Quality of Life, evaluated with EORTC-QLQ-C30
safety of EGCG | 12 month
  Number of adverse events according to CTC criteria (Version 4.0)
change in cardiac biomarkers | Baseline, 12 Month
  cardiac troponin T (hsTNT), NTproBNP
improvement of hematological remission | Baseline, 12 Month
  Hematological Response according to Palladini et al 2012
Organ response in affected organs other than heart | Baseline, 12 Month
  Organ response according to Gertz et al 2005
Overall Survival | 12 Month

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schönland, MD, Principal Investigator — University Hospital of Heidelberg
Locations (1):
- University Hospital of Heidelberg; Medical Department V, Heidelberg, Baden-Wurttemberg, Germany